CLINICAL TRIAL: NCT06823921
Title: Effects of High-Intensity Interval Training (HIIT) on Cognitive Function and Quality of Life in Parkinson's Disease: A Pilot Clinical Trial
Brief Title: Cognitive Effects of Exercise in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sule Tinaz (Other)
Responsible Party: Sponsor-Investigator, Sule Tinaz, Associate Professor of Neurology, Yale University
Organization: Yale University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000039232
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: exercise; high-intensity interval training; cognitive function; MRI
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Participants in the HIIT group will be expected to attend 3 exercise classes per week for 3 months
  Interventions: Other: Exercise
- Control (No Intervention): Participants in the control group will continue their standard care and usual physical activities

INTERVENTIONS:
Other: Exercise — HIIT will include aerobic, strength, and balance exercises and boxing
  Other Names: HIIT
  Arms: High-intensity interval training

SUMMARY:
This pilot study will evaluate the short-term (3 months) and long-term (6 months) effectiveness of a high-intensity interval training (HIIT) program in improving cognitive function and self-efficacy in individuals with PD.

DETAILED DESCRIPTION:
Participants will be assigned to either the HIIT group, which will engage in 3 classes per week, or a standard-of-care control group, which will include people who will continue their standard care and usual physical activities but do not plan on partaking in additional structured exercise interventions for 3 months (except for physical and occupational therapy if medically necessary). Cognitive functions will be measured using standardized tests (Stroop, Trail Making Test-B (TMT-B), verbal fluency (using letters F-A-S), and Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)), alongside assessing subjective ratings of daily cognitive function using the Neuro Quality of Life - Cognitive Function (Neuro-QoL CF) survey. Secondary outcomes will include self-efficacy measures, specifically regarding goal achievement, managing emotions and daily activities. We will also aim to obtain brain functional MRI (fMRI) and neuromelanin-sensitive MRI (NM-MRI) data from a subset of participants to measure the brain effects of HIIT as exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Age 40 year and above
* Willingness and ability to participate in HIIT exercise classes

Exclusion Criteria:

* Non-English speaking
* Neuropsychiatric disorder other than Parkinson's disease and comorbid depression and anxiety (e.g., stroke, epilepsy, brain tumor, multiple sclerosis, schizophrenia, bipolar disorder, obsessive compulsive disorder, etc.)
* High levels of exercise at baseline (exercising at high intensity at least 3 times per week or moderate intensity at least 5 times per week)
* Hoehn & Yahr disease stage > 3 (physically not independent)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Neurological Disorders (Neuro-QoL) cognitive function survey | 3 months and 6 months
  Subjective measures of cognitive functioning in daily life. It captures aspects of cognitive functioning such as attention, memory, and executive function. The average T-score is 50. Higher score indicates better performance.

SECONDARY OUTCOMES:
Executive function composite T-score | 3 months and 6 months
  Average T-scores of Trail Making Test-B, Stroop, and F-A-S verbal fluency test that are used to test executive functions. The average T-score is 50. Higher score indicates better performance.
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) memory domain index score | 3 months and 6 months
  Examines verbal and visual memory performance and calculates an index score (range: 40-160). Higher score indicates better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
This is an early-phase pilot study to determine feasibility.

REFERENCES:
- [Result] de Laat B, Hoye J, Stanley G, Hespeler M, Ligi J, Mohan V, Wooten DW, Zhang X, Nguyen TD, Key J, Colonna G, Huang Y, Nabulsi N, Patel A, Matuskey D, Morris ED, Tinaz S. Intense exercise increases dopamine transporter and neuromelanin concentrations in the substantia nigra in Parkinson's disease. NPJ Parkinsons Dis. 2024 Feb 9;10(1):34. doi: 10.1038/s41531-024-00641-1. PMID 38336768